CLINICAL TRIAL: NCT03575208
Title: Use of Hepatitis B Immune Globulin (HBIg) to Restore Immune Control in Patients With Chronic Hepatitis B
Brief Title: Hepatitis B Immune Globulin (HBIg) to Restore Immune Control in People With Chronic Hepatitis B
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow/Insufficient accrual
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180116; 18-DK-0116
Record Dates: First submitted 2018-06-29; First posted 2018-07-02 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Chronic Hepatitis B
Keywords: HBsAg Loss; Peginterferon; Inactive Carrier
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — hepatitis B hyperimmune globulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HBIG followed by Peginterferon alfa-2a (Experimental): HBIg x 12 weeks followed by peginterferon alfa-2a 180mcg x 24 weeks
  Interventions: Biological: hepatitis B immune globulin (HBIg); Drug: Pegylated interferon alfa (pegIFN)
- Peginterferon alfa-2a (Active Comparator): Peginterferon alfa-2a 180mcg x 24 weeks
  Interventions: Drug: Pegylated interferon alfa (pegIFN)

INTERVENTIONS:
Biological: hepatitis B immune globulin (HBIg) — HBIg 20,000 U/L iv. Dosing interval will depend on anti-HBs levels.
  Arms: HBIG followed by Peginterferon alfa-2a
Drug: Pegylated interferon alfa (pegIFN) — peginterferon alfa-2a 180 mcg weekly for 24 weeks

SUMMARY:
Background:

Hepatitis B is a viral infection of the liver. When the immune system tries to clear hepatitis B, it damages the liver. Eventually, the immune system gets exhausted fighting the virus. Researchers want to see if giving large doses of an antibody (HBIg) with the drug peginterferon will boost the immune system in people with this disease.

Objectives:

To observe the effect of large doses of antibody against the hepatitis B surface antigen on the immune response to the virus. To see if removing hepatitis B surface antigen from the blood enhances the action of peginterferon.

Eligibility:

Adults ages 18 and older with hepatitis B

Design:

Participants will be screened twice with a medical history, physical exam, and blood and urine tests.

Participants will be randomly put in one of two groups. All participants will get peginterferon for 24 weeks. One group will first get HBIg for 12 weeks.

Participants in the combination group will have a 4-day clinic stay. They will have:

Repeats of screening tests

Eye exam

Liver ultrasound

The first dose of HBIg by IV over 2 hours

These participants will get HBIg at the clinic up to 8 times over 12 weeks then start the peginterferon.

All participants will get peginterferon for 24 weeks. They will get it by injection under the skin once a week. They may do this themselves. They will keep a drug diary. They will have 5 visits to assess response and monitoring for safety..

After stopping the study drug, participants will have 4 follow-up visits over 36 weeks. They will repeat screening tests and have 1 liver ultrasound.

DETAILED DESCRIPTION:
Up to 300 subjects with hepatitis B e antigen (HBeAg) negative chronic hepatitis B who are inactive carriers (specified as those with HBV DNA levels <2,000 IU/mL over a 6-month period with ALT levels <1.5 X upper limit of normal and HBsAg level <1500 IU/mL) will be screened and 25 enrolled in a randomized trial of hepatitis B immune globulin (HBIg) for 12 weeks followed by peginterferon alfa for 24 weeks versus peginterferon alfa-2a alone for 24 weeks. The focus of the study is to understand mechanistically what effect the removal of HBsAg will have on the immune response and action of peginterferon alfa-2a. Chronic hepatitis B is characterized by immune exhaustion, which is felt to be caused by ongoing exposure of immune cells to high levels of viral antigens such as HBsAg. Presence of viral antigen results in continuous immune cell stimulation leading to functional exhaustion and progressive loss of immune function. In this study, we will attempt to achieve elimination of circulating HBsAg from the blood of chronically infected patients by administering high doses of hepatitis B immunoglobulin followed by peginterferon alfa-2a. A control arm consisting of peginterferon alfa-2a alone will be included to allow for assessment of the effect of HBIg on response to peginterferon alfa-2a. We will investigate whether this strategy will result in restoration of and/or increase in innate immunity leading to HBsAg clearance and development of long-lasting protective immunity. The proposed study will be conducted in three phases with pre-specified stopping rules to ensure subjects are responding appropriately at the end of each phase before moving to the next phase. The primary endpoints of the trial will be restoration of HBV-specific adaptive immunity at two time points (the end of HBIg treatment (week 12) and at the end of treatment (week 36) and increase in innate immune response to peginterferon alfa-2a treatment and a secondary endpoint will be a greater than 0.5 log10 reduction in HBsAg level at the study end point (week 36).

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Male or female >=18 years of age
* Known serum HBsAg positive with a level <1,500 IU/mL measured within 144 weeks of screening
* Hepatitis B e antigen negative at the time of screening
* HBV DNA levels <2000 IU/mL measured on two occasions at least 24 weeks and no more than 48 weeks apart, during screening
* ALT level <=1.5 ULN measured on two occasions at least 24 weeks and no more than 48 weeks apart, during screening

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Any treatment for HBV within the last 48 weeks
* Co-infection with HDV as defined by the presence of anti-HDV
* Co-infection with HCV as defined by the presence of anti-HCV with HCV RNA
* Co-infection with HIV as defined by the presence of anti-HIV
* Presence of anti-HBs
* Cirrhosis either diagnosed by a prior liver biopsy at any time or if not available by a transient elastography score >13 kPa.
* Decompensated liver disease as defined by serum bilirubin >2.5 mg/dL (with direct bilirubin > 0.5 mg/dL), prothrombin time of greater than 2 seconds prolonged, a serum albumin of less than 3.5 g/dL, or a history of ascites, variceal bleeding or hepatic encephalopathy.
* Presence of other causes of liver disease, (i.e. hemochromatosis, Wilson disease, alcoholic liver disease, alpha-1-anti-trypsin deficiency).
* A history of organ transplantation, or in the absence of organ transplantation any medical condition requiring the chronic use of more than 5 mg of prednisone (or its equivalent) daily.
* Severe IgA deficiency
* Severe allergic reaction to any human immunoglobulin product
* Significant systemic illness other than liver diseases including congestive heart failure, renal failure, chronic pancreatitis, and diabetes mellitus with poor control, that in the opinion of the investigator may interfere with therapy.
* Pregnancy or for women of childbearing potential, inability or unwillingness to use an effective form of contraception during study participation.
* Lactating women.
* Hepatocellular carcinoma (HCC), or the presence of a mass on imaging studies of the liver that is suggestive of HCC, or an alpha-fetoprotein level of greater than 500 ng/mL
* eGFR < 50 ml/min, serum creatinine > 1.3 mg/dL
* History of hypersensitivity to pegylated interferon-alpha
* Platelet count <90 mm3/dL
* Hgb <12 g/dL for males and <11 g/dL for females
* Active ethanol/drug abuse/psychiatric problems such as major depression, schizophrenia, bipolar illness, obsessive-compulsive disorder, severe anxiety, or personality disorder that, in the investigator s opinion, might interfere with participation in the study.
* History of malignancy or treatment for a malignancy within the past 3 years (except adequately treated carcinoma in situ or basal cell carcinoma of the skin).
* History of immune-mediated disease, or cerebrovascular, chronic pulmonary or cardiac disease associated with functional limitation, retinopathy, uncontrolled thyroid disease, poorly controlled diabetes or uncontrolled seizure disorder, as determined by a study physician.
* Presence of conditions that, in the opinion of the investigators, would not allow the patient to be followed in the current study.
* Inability of subject to understand and the unwillingness to sign a written informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
NK cell response to the first peginterferon injection both groups | 6 hours after the first peginterferon injection
  Change in TRAIL-expressing NK cell within the first 6 hours after the first peginterferon injection
Improvement of HBsAg-specific T cell responses HBIG only group | Baseline to week 12
  Change in the frequency of IFN-g producing T cells from baseline to week 12 as compared to HBV core and polymerase-specific T cell responses in the same patients
Improvement of HBsAg-specific T cell responses both groups | Baseline to week 36
  Change in the frequency of IFN-g producing T cells from baseline to week 36

SECONDARY OUTCOMES:
HBsAg loss | Up to week 84
  Loss of HBsAg confirmed on 2 consecutive visits at least 12 weeks apart at any time off therapy (HBIg and pegIFN)
Change in HBsAg from baseline to 48 weeks off peginterferon therapy | Week 84
  Change in log10 HBsAg from baseline to 48 weeks off peginterferon therapy
Change in HBsAg from baseline to 24 weeks off peginterferon therapy | Week 60
  Change in log10 HBsAg from baseline to 24 weeks off peginterferon therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Liu J, Yang HI, Lee MH, Lu SN, Jen CL, Batrla-Utermann R, Wang LY, You SL, Hsiao CK, Chen PJ, Chen CJ; R.E.V.E.A.L.-HBV Study Group. Spontaneous seroclearance of hepatitis B seromarkers and subsequent risk of hepatocellular carcinoma. Gut. 2014 Oct;63(10):1648-57. doi: 10.1136/gutjnl-2013-305785. Epub 2013 Nov 13. PMID 24225939
- [Background] Rehermann B. Pathogenesis of chronic viral hepatitis: differential roles of T cells and NK cells. Nat Med. 2013 Jul;19(7):859-68. doi: 10.1038/nm.3251. PMID 23836236
- [Background] Liang TJ, Block TM, McMahon BJ, Ghany MG, Urban S, Guo JT, Locarnini S, Zoulim F, Chang KM, Lok AS. Present and future therapies of hepatitis B: From discovery to cure. Hepatology. 2015 Dec;62(6):1893-908. doi: 10.1002/hep.28025. Epub 2015 Oct 27. PMID 26239691
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-DK-0116.html